CLINICAL TRIAL: NCT04034433
Title: Benefits of a Perioperative Exercise Program on Maturation of Dialysis Arteriovenous Fistulas
Brief Title: Exercise Program for Arteriovenous Fistula Maturation
Acronym: FAVULOUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 69HCL19_0215; ID-RCB (Other: 2019-A00767-50)
Record Dates: First submitted 2019-07-24; First posted 2019-07-26 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Arteriovenous Fistula
Keywords: Arteriovenous Fistula Diameter; Handgrip; Program exercise; Maturation
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise (Experimental)
  Interventions: Procedure: Handgrip exercise program
- Control (No Intervention)

INTERVENTIONS:
Procedure: Handgrip exercise program — Handgrip exercise with a rubber ball 4 weeks before the surgery until 4 weeks after the surgery 20 contractions per minute for a total of 20 minutes each day.
  Arms: Exercise

SUMMARY:
Arteriovenous fistula (AVF) is the recommended vascular access for chronic hemodialysis, as it is associated with less mortality and better patency than arteriovenous graft (AVG) or central venous catheter (CVC).

Unfortunately, AVF suffers from a high failure rate, due, in part, to poor venous diameter.

The aim of this study is to investigate whether a perioperative handgrip training can improve the diameter of AVF in patients with chronic kidney disease (CKD) (stage IV-V).

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* with chronic kidney disease (Estimated Glomerular Filtration Rate (eGFR) <30 milliLiter/minute (mL/min))
* with follow-up at the University Hospital of Lyon Sud
* who choose hemodialysis as renal replacement therapy

Exclusion Criteria:

* contraindication for arteriovenous fistula (AVF) surgery
* refusing AVF creation
* prior vascular access
* antecedent of IV substance abuse
* active cancer
* inability to perform handgrip exercise
* physical or mental disability limiting follow-up possibility
* inclusion in an other interventional study
* no social welfare

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-10-04 (Actual); Primary Completion 2026-11-04 (Estimated); Study Completion 2026-11-04 (Estimated)

PRIMARY OUTCOMES:
Arteriovenous Fistula (AVF diameter) | at 6 weeks (after surgery)
  Arteriovenous Fistula diameter will be measured by Doppler ultrasound

SECONDARY OUTCOMES:
Echographic maturation rate | at 6 weeks (after surgery)
  Maturation rate of Arteriovenous Fistula (AVF) by echography defined as blood flow>600milliLiters/minute (mL/min), diameter>6millimeters (mm) and depth <6mm
Clinical maturation rate | at 6 weeks (after surgery)
  Arteriovenous Fistula (AVF) measured by a vein easily palpable, relatively straight, with a uniform sensation of quivering and more than 10centimeters (cm) long.
Arteriovenous Fistula (AVF) localization (arm or forearm) | at 6 weeks (after surgery)
  After the patient's examination, the vascular surgeon will choose the future AVF localization
Arteriovenous Fistula (AVF) interventions | up to 6 weeks
  Necessity of performing an intervention (such as angioplasty or thrombolysis or thrombectomy or superficialization) on the Arteriovenous Fistula (AVF)
Emergency hemodialysis on Central Venous Catheter (CVC) | up to 6 weeks
  Necessity of patients on CVC to undergo emergency hemodialysis
Emergency hemodialysis on Arteriovenous Graft (AVG) | up to 6 weeks
  Necessity of patients on AVG to undergo emergency hemodialysis

CONTACTS AND LOCATIONS:
Overall Officials: Abbas DEEB, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Service de néphrologie, dialyse et nutrition rénale - Centre Hospitalier Lyon Sud, Pierre-Bénite, France